CLINICAL TRIAL: NCT01020851
Title: The PREVENTS Trial: The Preventing Recurrent Events in Veterans Navigating TIA or Stroke Trial
Brief Title: The PREVENTS Trial: The Preventing Recurrent Events in Veterans Navigating Transient Ischemic Attack (TIA) or Stroke Trial
Acronym: PREVENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Narrows Institute for Biomedical Research (Other)
Responsible Party: Principal Investigator, Jennifer Friedberg, Clinical Psychologist, Narrows Institute for Biomedical Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AHA0835195N
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Stroke; Transient Ischemic Attack
Keywords: hypertension; stroke; cholesterol; adherence
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Hypertension | interventions — Transtheoretical Model

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tailored intervention (Experimental): Participants in this arm will receive 6 monthly telephone calls of a behaviorally tailored intervention based on the transtheoretical model.
  Interventions: Behavioral: tailored intervention
- attention placebo (Active Comparator): Participants in this arm will receive 6 monthly telephone delivered counseling sessions about general health topics
  Interventions: Behavioral: attention placebo

INTERVENTIONS:
Behavioral: tailored intervention — 6 monthly telephone calls focusing on diet, medication and exercise adherence using the framework of the transtheoretical model
  Other Names: stage-matched intervention; transtheoretical model
  Arms: tailored intervention
Behavioral: attention placebo — 6 monthly telephone-delivered sessions focusing on general health topics
  Arms: attention placebo

SUMMARY:
National recommendations state that patients with a history of transient ischemic attack (TIA) or ischemic stroke should receive hypertension treatment, including antihypertensive medication and lifestyle modification, with a goal of reducing blood pressure (BP) to <120 mm Hg systolic BP and <80 mm Hg diastolic BP. Statin treatment and lifestyle modification is also recommended for post-stroke and post-TIA patients with elevated cholesterol levels or a history of stroke or TIA with an atherosclerotic cause. Despite the clear benefits of secondary stroke prevention, there is a gap between evidence and implementation in clinical practice. By a randomized controlled trial, the investigators will test whether a tailored, telephone-delivered transtheoretical model-based behavioral intervention will improve adherence to treatment in veterans with a history of TIA or stroke, thereby leading to better control of BP and cholesterol levels, as compared to an attention placebo.

The primary specific aims of this project are to:

* determine whether a behaviorally tailored intervention (TI) can effectively lower BP after 6 months of counseling as compared to an attention placebo (AP) in veterans with a history of stroke or TIA
* assess whether the TI is effective in improving adherence to diet after 6 months of counseling in veterans with a history of stroke or TIA.

Secondary aims are to

* assess whether the TI is effective in improving cholesterol levels in post-stroke veterans after 6 months
* evaluate whether the TI is effective in improving adherence to antihypertensive and lipid-lowering medications after 6 months of counseling in veterans with a history of stroke or TIA
* determine whether the TI is effective in improving adherence to exercise recommendations after 6 months.

To answer this, veterans (n=190) with a history of stroke or TIA will be randomized equally to the TI, which will use the transtheoretical framework to provide 6 monthly counseling phone sessions about adherence to diet, medication, and exercise recommendations, and the AP, in which 6 monthly counseling phone sessions about non-stroke-related health topics will be provided. Participants will make in-person visits at baseline and 6 months. BP (3 measures taken at least 5 min apart) and dietary sodium are the primary outcomes, while secondary outcomes will be total cholesterol/high density lipoprotein ratio, adherence to antihypertensive and lipid-lowering drugs, and exercise adherence.

ELIGIBILITY:
Inclusion Criteria:

* Well-documented history of stroke or TIA
* Age 21 years or older
* Continuity of care in the primary care or neurology clinics, defined as at least 1 visit in either clinic during the past 1 year
* On hypertensive and/or lipid-lowering agents
* A score of >16 on the Mini-Mental Status Exam-
* Ability to exercise (assessed by time to get up and go).

Exclusion Criteria

* Limited life expectancy due to a severe non-CVD related comorbid terminal illness such as cancer
* No telephone number at which patient can be reached
* Plans to relocate within the next 6 months
* Inability to communicate over the telephone due to severe cognitive impairment or aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2008-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
blood pressure | 6 months

SECONDARY OUTCOMES:
cholesterol | 6 months
dietary adherence | 6 months
exercise adherence | 6 months
medication adherence | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- VA New York Harbor Healthcare System, NY and Brooklyn Campuses, New York, New York, United States